CLINICAL TRIAL: NCT01615016
Title: Feasibility Study of A Comparison of Minimally Invasive Surfactant Application Techniques in Preterm Infants
Brief Title: MISurf Versus InSurE. A Comparison of Minimally Invasive Surfactant Application Techniques in Preterm Infants
Acronym: MIsurf
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Delay due to infrastructural reasons. Funding withdrawn
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, elhelous, Dr. med. / Associate Professor, Hamilton Health Sciences Corporation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: NIF-12295
Record Dates: First submitted 2012-05-30; First posted 2012-06-08 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Hyaline Membrane Disease
Keywords: Preterm infant; Surfactant application; Respiratory Distress Syndrome; Minimally invasive Surfactant Application; INSURE (Intubate-Surfactant-Extubate)
MeSH Terms: conditions — Hyaline Membrane Disease; Premature Birth; Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized, double blind
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Intervention team whose members are not part of the patients' care team. Blinded for type of intervention
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MISurf (Experimental): Minimally Surfactant application via small tube inserted into the trachea under CPAP therapy without formal intubation and without mechanical ventilation
  Interventions: Other: Minimally invasive endotracheal surfactant application
- InSurE (Active Comparator): Surfactant application via Intubation - Surfactant Application - Extubation sequence
  Interventions: Other: Minimally invasive endotracheal surfactant application

INTERVENTIONS:
Other: Minimally invasive endotracheal surfactant application — What are the planned trial interventions?
  1. MISurf: Minimally invasive intratracheal surfactant application without mechanical ventilation by feeding tube device
  2. InSurE: Surfactant application by InSurE strategy (Intubation - surfactant - extubation sequence).
  Both interventions will be performed by intervention teams. For the MISurf intervention, it was decided to use the minimally invasive method via feeding tube exclusively due to concerns about possibility of airway injury with the iv cannula device.
  Surfactant Two porcine derived surfactant products have been used in the published trials for minimal invasive surfactant application, Curosurf© and Survanta©. Due to safety reasons we will use these products also in our pilot study however, only the latter is currently available in Canada. Hence we will use Survanta© 100 mg/kgBW, equivalent to 4 ml/kgBW per dose.19,20,26
  Other Names: Surfactant Application via feeding tube.; Non invasive surfactant application.

SUMMARY:
The lungs of infants born too early are extremely underdeveloped. Respiratory Distress Syndrome (RDS) is a condition that frequently develops in infants born more than 10 weeks early and leads to the collapse of their lungs. Because the lungs had not had enough time to mature, they lack a substance, called surfactant that prevents their collapse. To treat this problem, physicians apply surfactant to the lungs within the first few hours of life by way of the infant's airway using mechanical stimulation (ventilation). Although this treatment has significantly decreased the number of infants who die from RDS, the mechanical ventilation can cause damage to the tiny lungs that may lead to long term lung disease and breathing problems.

The need for more gentle and less invasive methods of deliver the surfactant to the infant has led to the development of two new methods that require little or no mechanical ventilation. While both methods are known to work there is no study that has assessed whether one method is better than the other or causes fewer complications for the infant. The proposed study will determine if it is practical to conduct a clinical trial to compare both methods of surfactant administration and to gather preliminary data on which method gives better results. Should this study look promising, the resulting data will be used to design a larger clinical trial to compare the methods of mechanical ventilation. Results of such a trial would help us to understand the best way to administer surfactant to preterm infants and thus help doctors to better care for tiny infants at risk of lung disease.

DETAILED DESCRIPTION:
1. The Need for a Trial What is the problem to be addressed? Respiratory distress syndrome (RDS) is a major clinical challenge affecting 60% of babies born before 30 weeks gestation and significantly contributes to mortality and morbidity in very preterm infants, including chronic lung disease and bronchopulmonary dysplasia. Given that the immature lungs of these tiny infants are developmentally deficient in surfactant, exogenous surfactant administration might be beneficial to prevent pulmonary atelectasis. The traditional method in preterm infants is via endotracheal tube accompanied by mechanical ventilation using positive pressure. The latter predisposes to permanent lung injury.This study seeks to assess the feasibility of conducting a large-scale clinical trial to compare two minimally invasive methods of surfactant administration to very low birth weight preterm infants. As such a comparative study has not been reported, the proposed study is a pilot trial to test the feasibility of the study design and to gather preliminary data on the comparison of two methods of surfactant administration. Results from this study will inform the design of a larger clinical trial including appropriate power calculation.

   Current management of lung disease in preterm infants RDS significantly contributes to mortality and morbidity in very preterm infants and is, itself, a major determinant of chronic lung disease (CLD) in the premature infant. One of the most common causes of RDS is surfactant deficiency; therefore, exogenous surfactant is frequently used for the treatment of RDS of the preterm infant. Endogenous surfactant is typically produced by alveolar cells type II and this substance, among other functions, decreases and modulates the surface tension in the small gas exchanging units of the lung, the alveoli.1 It has been shown that surfactant treatment is more effective when used within first hours of life rather than later as rescue therapy. The traditional method of surfactant administration is via an endotracheal tube where the infant is intubated and mechanically ventilated, with the latter often resulting in a pulmonary inflammatory response. This response is known to be a significant contributor to the development of CLD which is the main pulmonary morbidity, both in the short and long term, associated with premature birth, thus traditionally supporting the need for mechanical ventilation in a highly vulnerable phase of lung development. Despite advances in management of respiratory distress, about 30% of infants born under < 1,000 g still develop CLD - defined as an oxygen need at 36 weeks postmenstrual age. Some of these infants develop severe lung disease requiring ventilation and/or supplemental oxygen for months or years. Significant contributors to this adverse long term outcome of premature birth are oxidant - and ventilation mediated injury and inflammation, leading to disrupted alveolarization and septation of the lungs.

   One well established therapy to prevent RDS is antenatal administration of steroids to mothers with imminent preterm birth for induction of lung maturation, a treatment that has resulted in significant improved outcome following preterm birth. This treatment results in improved neonatal lung compliance with fewer infants requiring exogenous surfactant therapy.7 The increasing use of this intervention has led to more infants not necessarily requiring postnatal surfactant and thus reduced need for mechanical ventilation, which allows to manage even extreme low birth weight infants with non-invasive pressure support as CPAP (continuous positive airway pressure) to establish functional residual capacity.

   Postnatal non-invasive respiratory support using continuous positive airway pressure (CPAP) has been shown to be effective in reducing lung damage in several studies, especially when initiated during the immediate postnatal adaptation period. This results in fewer days of ventilation and a trend towards a lower risk of CLD, when compared to intubated and mechanically ventilated controls. However, the number of infants who are started on CPAP but who ultimately require intubation for the administration of exogenous surfactant within the first 72 hours remains high in the extremely low birth weight category. Usually CPAP failure is due to unremitting RDS requiring surfactant therapy. There is evidence that failing CPAP therapy, defined as need for intubation within 72 hours of postnatal age, is associated with adverse outcome in infants between 25 to 28 weeks gestation with a higher risk of CLD, death or CLD and necrotizing enterocolitis. In the same trial infants between 29 and 32 weeks of gestation failing CPAP were at higher risk of pneumothorax.

   In current clinical practice neonatologists are faced with the quandary of avoiding mechanical positive pressure ventilation, but with the knowledge that surfactant treatment is more effective in earlier phases of RDS, and that CPAP failure could lead to higher risk of an adverse outcome. Hence efforts have been made to develop non-invasive strategies of surfactant application to take advantage of the high efficacy of this treatment and to decrease duration of mechanical ventilation and subsequent lung injury. To date, all attempts to produce an effective surfactant for nebulization have been unsuccessful.

   Recent advances in treatment of RDS In 1999, a Swedish group developed the InSurE procedure of surfactant administration, which involves intubation solely for the purpose of surfactant administration followed by immediate extubation to CPAP, thereby avoiding prolonged positive pressure ventilation. A Cochrane systematic review in 2008 concluded that this method, when compared with later selective surfactant therapy and continued mechanical ventilation, is associated with less need for mechanical ventilation, lower incidence of CLD and fewer air leak syndromes. InSurE has been shown to be effective even if used multiple times in the same patient. Failure of InSurE was associated with severity of RDS and extremely low birth weight < 750g. The CURPAP trial compared prophylactic administration of surfactant using the INSURE technique with early CPAP and early selective surfactant therapy if required. This trial found no difference for the outcome of mechanical ventilation in the first 5 days of life.

   Minimally invasive surfactant application (MISurf) via feeding tube or IV cannula device is a recently described innovative method of surfactant administration without the need for positive pressure ventilation. Using the same technique of visualization of the larynx by direct laryngoscopy as with classical intubation, the respective device is positioned in the infant's trachea, surfactant is applied, and the device is removed immediately without mechanical ventilation; If not already on CPAP, the patient is placed on nasal CPAP immediately following the procedure. In a large open-label multi- center randomized controlled trial, this method significantly reduced the need for mechanical ventilation in preterm infants between 26 and 28 weeks of gestation.

   What is/are the principal research question(s) to be addressed? This pilot study seeks to assess the feasibility of conducting a large-scale randomized trial to compare the two described methods of delivering surfactant, MISURF and INSURE. If this study design proves feasible, a larger trial would test the hypothesis that early surfactant administration via feeding tube/ IV cannula device under complete avoidance of mechanical ventilation as compared to INSURE will decrease the incidence and duration of invasive ventilation in the whole study population and decrease the incidence of CLD in infants of 25-28 week gestation.

   Why is a trial needed now? Evidence shows that the classical, invasive way of administering surfactant therapy is associated with serious side effects. This method is currently the most commonly used in neonatology, including at McMaster. MISurf and InSurE are the most common minimally invasive surfactant application techniques used in neonatology; InSurE is considered best practice for minimally invasive application and MISurf is promising practice. They have been compared to either CPAP therapy or to the classical way of administering surfactant with some evidence of benefit. No systematic review exists of randomized trials using minimally invasive surfactant delivery. Our literature review with search terms of surfactant therapy, minimal invasive surfactant application, InSurE, comparison, preterm infant, non invasive surfactant application, in different combinations, has not revealed one trial comparing these two methods directly with each other. The combination of minimally invasive surfactant application without mechanical ventilation with early CPAP therapy should offer the best lung protective strategy. A theoretical counter-argument could be that administering surfactant without the pressure of the ventilation (MISurf), the distribution of surfactant into the lung tissue could be less efficient compared to (INSurE) where intubation and surfactant administration are accompanied by positive pressure ventilation. Hence a comparative randomized trial will significantly contribute to the evidence and knowledge about the role of these two minimal invasive strategies for surfactant administration and as such influence or respectively change practice at Hamilton Health Sciences and beyond. The outcome of this trial could support the rationale for a multicenter trial throughout Canada.

   Why is a pilot study necessary? As this will be the first study to compare these two methods, aspects of feasibility have to be tested. The design of the proposed pilot study is a randomized, two armed intervention trial, with a masked intervention. It is vital to investigate if the procedures of the trial and masking of intervention are feasible. Recruitment rate, drop-out rate because of meeting exclusion criteria, refusal rate, consent- and randomization process, acceptance by clinicians and staff, also need to be investigated. The results of this pilot trial will inform the sample size calculation of a larger trial. This pilot will also confirm acceptability of study inclusion criteria.

   Clinical relevance As described above, CPAP therapy alone might lead to unfavorable outcome in a group of patients using intubation failing this treatment and needing rescue surfactant therapy. However, undertaking surfactant therapy in all extreme premature infants is not considered good clinical practice. What is needed is to be able to identify the patient group who is most likely to benefit from surfactant therapy, and then to define the optimal time and method of surfactant application. This should lead to better outcome due to less days of ventilatory treatment, translating in significant decrease of cost in the short term (one surfactant application costs between 300 to >1000$, depending on product and country) as well as long term, considering the burden costs of CLD, with children needing specialist care for the first years of life.
2. The Proposed Trial

   Study Design We propose to assess the feasibility of a masked, prospective randomized controlled trial, with two intervention arms, to compare surfactant application using the InSurE technique versus the MISurf technique. As early CPAP therapy is currently the standard of care for patients less than 33 weeks gestation, patients in both arms of the study will receive this intervention.

   What are the planned trial interventions?
   1. MISurf: Minimally invasive intratracheal surfactant application without mechanical ventilation by feeding tube device
   2. InSurE: Surfactant application by InSurE strategy (Intubation - surfactant - extubation sequence).

   Both interventions will be performed by intervention teams, comprised of an attending physician, a neonatal fellow, a respiratory therapist, nurse practitioner and nurses. The physical visualization and application of surfactant will be performed by the attending physician or the neonatal fellow, who is part of the intervention team. For the MISurf intervention, it was decided to use the minimally invasive method via feeding tube exclusively due to concerns about possibility of airway injury with the iv cannula device.

   Surfactant Two porcine derived surfactant products have been used in the published trials for minimal invasive surfactant application, Curosurf© and Survanta©. Due to safety reasons we will use these products also in our pilot study however, only the latter is currently available in Canada. Hence we will use Survanta© 100 mg/kgBW, equivalent to 4 ml/kgBW per dose.

   Medication Considering the non invasiveness of the procedure, medication (anaesthetic agents, analgosedation) will not be administered for study interventions.

   What are the proposed practical arrangements for allocating participants to trial groups? This pilot trial will allocate participants to groups using simple randomization with sealed nontransparent envelopes. Every eligible patient for whom parental consent has been obtained will be randomized after birth.

   What are the proposed methods for protecting against sources of bias?

   Details of masking procedure Intervention teams will be established and will be comprised of health professionals (as above) who are not part of the infants' care team within the first 3 days of life. The procedure itself will be performed either in a different room (infant stabilization room (ISR)), or behind a folding screen.

   Blinding of health professionals in the circle of care Eligible patients will be randomized at birth or as soon thereafter as possible, once parental consent has been obtained. Professionals in the infant's circle of care and those assessing outcome will be blind to their study group.

   What are the planned inclusion/exclusion criteria? Eligible are all preterm infants born ≤ 30 weeks gestation at McMaster Inclusion criteria
   * CPAP of 5-6 cm H2O and FiO2≥ 0.35 or CPAP of 7-8 cm of H2O and FiO2≥ 0.30
   * Less than 36 hours of age
   * Worsening clinical signs of RDS such as retractions (clinical judgment of the responsible physician) Exclusion Criteria
   * Previous Intubation or in imminent need of invasive mechanical ventilation because of e.g. apnea, severe bradycardia or other deterioration not attributed to RDS, e.g. shock
   * Congenital anomaly or conditions that might adversely affect breathing
   * Pneumothorax before intervention
   * No parental consent

   What is the proposed duration of treatment period? Infants are eligible to enter the study for intervention within 36h of life. The intervention itself will take 5 to 15 minutes. A second (one repeat) non invasive intervention is allowed in case of a second surfactant dose to be required.

   What is the proposed frequency and duration of follow up? Outcome will be assessed within first 3 days of life, within 48 hours after intervention and until discharge.

   What are the proposed primary and secondary outcome measures?
3. Primary feasibility outcome

   • Proportion of included infants who were treated according to protocol
4. Secondary feasibility outcome

   * Recruitment rate
   * Consent rate
   * Proportion of intervention procedures in which masking has not been successful
   * Proportion of interventions, when intervention team has not arrived in time leading to emergency intervention
   * Success rate in antenatal approach for consent
5. Primary clinical outcome

   Failure rate of the intervention, where failure is defined as:
   * Need for invasive ventilation, requiring either FiO2 more than 0.6 or pCO2 more than 65 mm Hg and pH < 7.20 or both for more than 2 hours after surfactant administration up to 72 hrs of life
   * Intubation/requirement for mechanical ventilation within 48h after first intervention (same criteria as above)
   * For InSurE: Failed extubation within 15 min after intubation for surfactant application
   * SAE during immediate intervention leading to intubation (e.g. severe bradycardia/resuscitation, pneumothorax)
6. Secondary clinical outcome

   * Proportion of infants not requiring the intervention
   * Proportion of the following co-morbidities until discharge? - Incidence of grade 3 and 4 IVH (intraventricular hemorrhage), - PVL (periventricular leucomalacia), - ROP (retinopathy of prematurity) requiring treatment, - NEC (necrotizing enterocolitis) stage 2 and 3
   * Total duration of invasive and non-invasive ventilation (extubation criteria will follow the extubation- and weaning guidelines), duration of oxygen supplementation until discharge
   * Proportion of patients requiring oxygen supplementation at discharge
   * Proportion of surfactant related adverse events like tube blockade, episodes of desaturation, bradycardia, pulmonary hemorrhage, pneumothorax differ in the two groups
   * Total number of surfactant doses required compared in the two groups
   * Incidence of CLD. CLD is assessed as per physiological CLD definition with the severity score of mild, moderate and severe
   * Death

   How will the outcome measures be measured at follow up? Clinical outcome data will be collected from patient medical records by the research coordinator and verified by the principal investigator. Feasibility outcome data will be documented by the intervention teams and collected by the research coordinator.

   What are the criteria for success of this pilot study? We aim to verify that it will be possible to perform a large scale clinical trial with this study design. Given that currently almost 100% of our patients are treated with classical surfactant application, a rate of >50 % of recruited patients treated according to protocol and a recruitment and consent rate indicating that a large scale trial with a estimated sample size of 150 to 200 patients within 2 to 3 years can be performed will determine success of this pilot trial.

   Sample size

   The sample size was primarily determined based on feasibility considerations. To test the feasibility of the study design a total of 40 patients (that is, 20 patients in each arm).In general, we estimate that 200 preterm infants are admitted to McMaster NICU per year and 40% of these would fulfill the eligibility criteria for this trial. Thus, we will have sufficient numbers to assess the feasibility of recruitment for the main trial. Main study:

   The sample size will be calculated based on results of the pilot study.

   What is the planned recruitment rate? How will the recruitment be organized? Over what time period will recruitment take place? What evidence is there that the planned recruitment rate is achievable? Where possible, recruitment will take place antenatally. The research coordinator will screen the Labour & Delivery high risk patients for eligibility. Mothers will then be informed of the study and approached for consent, if they provide consent to contact. A recruitment rate of more than 70% should be achievable based on previous experience with clinical studies in our unit with this population. All infants of gestational age < 30 weeks are eligible. Based on the data for McMaster NICU from Vermont Oxford Network and Canadian Neonatal Network around a proportion of 40% of these patients is estimated to meet the inclusion criteria for the intervention.

   What is the proposed type of analyses? The reporting of this pilot trial will be in accordance with the CONSORT Statement (www.consort-statement.org). The demographics and baseline characteristics of the trial participant will be analyzed using descriptive statistics reported as mean standard deviation [SD] or median (minimum, maximum) for continuous variables depending on the distribution, and count (percent) for categorical variables. The feasibility outcomes will be reported as percentages. For clinical outcomes, we will use the t-test for comparing groups on continuous outcomes and chi-squared test for categorical variables. All tests will be performed at alpha = 0.05 level of significance. We will not adjust the overall level of significance for multiple testing as the tests will be primarily exploratory. All analyses will be performed using SAS 9.2 (Cary. NC).

   What is the proposed frequency of analyses? Interim analysis will be conducted following inclusion of first 20 patients, which is expected at around 6 months, under the assumption of a population of 200/year, recruitment rate of 70% and an eligibility rate for entering one of the intervention arms of 40%.

   Safety DSMB: Considering the patient population and the intervention a DSMB will be established. This will comprise of an external trialist/statistician, an external neonatologist and an external experienced clinical researcher outside the subject area. SAEs: SAEs will be captured and reported to DSMB within 24h.

   Alternative treatment: There is a considerable amount of patients (around 25%) who will not require intervention and will remain on CPAP treatment alone.31 The alternative pathway would be intubation and mechanical ventilation due to various causes of respiratory failure.

   Ethical considerations Full approval of the FHS/HHS REB will be obtained prior to commencement.
7. Risks to the safety of participants involved in the trial Although this is the first time these interventions have been compared neither intervention is considered technically challenging or new. Hence no enhanced risk compared to the classical surfactant application is expected. The thresholds for intervention are chosen according to best practice recommendations and similar to other surfactant trials.14-21,26,28,29 Adverse events related to the intervention such as pneumothorax, tube blockage, pulmonary hemorrhage will be treated with current best practice intensive care as any other complication. They will be reported as described under 2.15.
8. Informed consent Written informed parental consent will be obtained by the research coordinator or by a physician who is not involved in the intervention team or the infant immediate care, when the coordinator is not available. Efforts will be undertaken to obtain parental consent prenatally. This should be feasible in most cases as more than 80% of the women with imminent preterm birth receive an antenatal consult by Neonatology and can be informed about the study at that point. When antenatal consent is not possible, consent will be taken as soon as achievable after birth, if the infant meets eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

Eligible are all preterm infants born ≤ 30 weeks gestation at McMaster Inclusion criteria

* CPAP of 5-6 cm H2O and FiO2≥ 0.35 or CPAP of 7-8 cm of H2O and FiO2≥ 0.30.21,22,26
* Less than 36 hours of age
* Worsening clinical signs of RDS such as retractions (clinical judgment of the responsible physician)

Exclusion Criteria:

* Previous Intubation or in imminent need of invasive mechanical ventilation because of e.g. apnea, severe bradycardia or other deterioration not attributed to RDS, e.g. shock
* Congenital anomaly or conditions that might adversely affect breathing
* Pneumothorax before intervention
* No parental consent

Max Age: 36 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2012-07; Primary Completion 2017-08-19 (Actual); Study Completion 2017-08-19 (Actual)

PRIMARY OUTCOMES:
Proportion of included infants who were treated according to protocol | Feasibility criteria endpoint after 12 months

SECONDARY OUTCOMES:
Recruitment rate | 1 year.
  * Recruitment rate
  * Consent rate
  * Proportion of intervention procedures in which masking has not been successful
  * Proportion of interventions, when intervention team has not arrived in time leading to emergency intervention
  * Success rate in antenatal approach for consent

CONTACTS AND LOCATIONS:
Overall Officials: Salhab el Helou, MD/AssocProf, Principal Investigator — McMaster University Children's Hospital/Hamilton Health Sciences
Locations (1):
- McMaster University Children's Hospital, Hamilton, Ontario, Canada